CLINICAL TRIAL: NCT04602130
Title: The Effect of Massage, Wipe Bathing and Tub Bathing on Physiological Measurements of Late Premature Newborns: A Randomised Controlled Trial
Brief Title: The Effect of Massage, Wipe Bathing and Tub Bathing on Physiological Measurements of Late Premature Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Yeliz SUNA DAĞ, Principal Investigator, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Yaşam bulgusu
Record Dates: First submitted 2020-09-17; First posted 2020-10-26 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Premature Newborn; Nurse; Physiological Measurements
MeSH Terms: conditions — Premature Birth | interventions — Control Groups; Massage

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Massage (Experimental): Massages were performed starting from the face, focused on the newborns forehead, and then around the eyes and cheeks with gentle touches. Then, newborns' chest area and the upper and lower extremities were massaged. Finally, newborns'were placed prone position and the back was massaged. Nurses recorded newborns' physiological measurements (pulse, respiration, oxygen saturation and body temperature) on the Newborn Follow-up Form.
  Interventions: Other: Control; Other: Sponge Bathing; Other: Tub Bathing
- Sponge Bathing (Experimental): In the sponge bathing group, the newborns' eyes, faces (outward from the midline), around the ear and the back of the ear were wiped from the inside out with cotton wipes and dried. Then, the chest area and arms, abdomen and back, legs and feet, respectively, were wiped and dried. Finally, the genital area was cleaned, before diapering the newborn. Nurses recorded newborns' physiological measurements (pulse, respiration, oxygen saturation and body temperature) on the Newborn Follow-up Form
  Interventions: Other: Control; Other: Massage; Other: Tub Bathing
- Tub bathing (Experimental): In the tub bathing group, before being immersed in the tub, the newborns' faces and heads were cleaned outwards from the midline and dried. Then, the neck, chest, arms, back, legs and genital area were soaped, before the full body was rinsed and dried. Finally, umbilical cord care was performed, and the baby was diapered. Nurses recorded the newborns' physiological measurements (pulse, respiration, oxygen saturation and body temperature) on the Newborn Follow-up Form.
  Interventions: Other: Control; Other: Massage; Other: Sponge Bathing
- Control (No Intervention): The newborns in the control group did not undergo any intervention other than standard clinical practices. All physiological measurements (pulse, respiration, oxygen saturation and body temperature) were performed by nurses and recorded on the Newborn Follow-up Form.

INTERVENTIONS:
Other: Control — The control group (n: 48) received no intervention except for the routine clinical practices. The newborns' physiological measurements before, immediately after and 30 minutes after the interventions were taken and recorded on the "Newborn Follow-up Form."
  Other Names: Control Group
  Arms: Massage; Sponge Bathing; Tub bathing
Other: Massage — The researcher applied massage (n: 48) to the newborns. The newborns' physiological measurements before, immediately after and 30 minutes after the interventions were taken and recorded on the "Newborn Follow-up Form."
  Other Names: Massage Group
  Arms: Sponge Bathing; Tub bathing
Other: Sponge Bathing — The researcher applied sponge bathing (n: 48) to the newborns. The newborns' physiological measurements before, immediately after and 30 minutes after the interventions were taken and recorded on the "Newborn Follow-up Form."
  Other Names: Sponge Bathing Group
  Arms: Massage; Tub bathing
Other: Tub Bathing — The researcher applied tub bathing (n: 48) to the newborns. The newborns' physiological measurements before, immediately after and 30 minutes after the interventions were taken and recorded on the "Newborn Follow-up Form."
  Other Names: Tub Bathing Group
  Arms: Massage; Sponge Bathing

SUMMARY:
Purpose: This randomized experimental study aimed to analyze the effect of massage, wipe bathing and tub bathing of late premature newborns on their physiological measurements.

Design and Methods: . This randomized experimental study was conducted on 192 newborns at the gestational week of 34 or higher in the newborn intensive care unit of a university hospital. The researcher applied massage (n: 48), tub bathing (n: 48), and wipe bathing (n: 48) to the newborns. The control group (n: 48) received no intervention except for the routine clinical practices. The newborns' physiological measurements before, immediately after and 30 minutes after the interventions were taken and recorded on the "Newborn Follow-up Form." The statistical analysis was performed using percentages, means, and ANOVA test.

DETAILED DESCRIPTION:
The neonatal period covers the postnatal first 28 days. During this period, newborns try to adapt to the extrauterine life after the intrauterine life and stabilize their respiratory and circulatory functions. Therefore, the acquisition of information on newborns' vital signs is crucial in the evaluation of and caregiving for newborns. The increase in evidence-based studies in nursing has led to changes and developments in the caregiving instructions that have hitherto been used in newborn intensive care units. However, the required and effective nursing practices that are considered indispensable in newborn intensive care units may cause various physiological (increase or decrease in heart and respiration rate, temporary decrease in oxygen saturation, hypothermia) and behavioral reactions (crying, uneasiness) Nurses, therefore, should closely monitor newborns' vital signs and make various interventions to keep these signs within normal values, as a primary practice.

The literature includes many studies conducted by nurses that focus on keeping newborns' physiological measurements within normal values. Massage means the stimulation of the soft tissues in the body. Previous studies have indicated that massage has positive effects such as relaxing the muscles, relieving pain, reducing bilirubin values by enabling blood and lymphatic circulation, increasing sleep duration, and strengthening the relationship between mothers and newborns. However, only a limited number of studies exist on the effects of massage on newborns' physiological measurements reported that the tactile stimulus through massages supported premature infants' parasympathetic functions and positively affected the infants' heart rate by reducing neurochemical and stress stimuli. Furthermore, Dieogo et al. (2008) reported that premature infants' body temperature increased due to the increased blood circulation during massage.

The bathing of newborns plays a highly important role in routine newborn clinical care practices, as well as in the individual, aesthetic, cultural, and hygienic benefits it confers. In neonatal intensive care units (NICU), tub baths, wipe baths, swaddle baths and shower-type bathing are commonly used. In Turkey, however, wipe baths and tub baths are often the most commonly used bathing methods in neonatal intensive care units . Although the literature shows differences among the institutions and countries, in newborn care units, wipe bathing is generally carried out by nurses, and tub bathing is not recommended until the infants' naval cord falls of. Numerous studies have shown that bathing can be performed without harming the newborn. Bryanton et al. (2004) indicated in their study that thermoregulation was ensured for the infants by drying them under a radiant warmer and placing them in an incubator. Mörelus et al. (2006) reported that infants might show physiological reactions, such as increased respiration and heart rate, to any stress. They also found that bathing positively affected infants' physiological measurements by relaxing them and reducing their stress levels. Studies that compare the effects of traditional wipe and tub bathing on newborns' physiological measurements have shown that tub bathing had more positive effects than wipe bathing. However, no studies have analyzed in the related literature that investigate the effects of massage, wipe bathing and tub bathing on physiological measurements, in the studies also have several inconsistencies, such as a small sample size, the failure to use control groups and a lack of blinding and follow-up. This randomized experimental study aimed to analyze the effect of massage, wipe bathing and tub bathing of late premature newborns on their physiological measurements.

Study design, setting, and population This study was conducted as a randomised controlled study between January and December 2018 in the NICU of a university hospital in Turkey. The NICU employs 30 nurses who provide newborns with bathing care performed routinely between 2 and 3 pm each afternoon.

In this study, permission to conduct the research was obtained from the hospital and the Inonu University Health Sciences Scientific Research and Publication Ethics Committee. All parents who agreed to participate in the research were informed of its methods and purpose, and each completed an informed consent form.

The study sample included the newborns who a) were born at 34 weeks' gestation and over b) were receiving routine care and who were stable (temperature >36.5 °C, SpO2> 95%, HR = 120-160 / min) c) had an apgar score of 7 or higher at the first minute after birth; d) were at least 24 hours old and who had no health problems that prevent bathing (e.g., congenital anomaly, surgical intervention, etc.) were included in the research.

The G*Power software package was used to calculate the sample size. The sample consisted of 192 newborns who comprised (d=0.5)effect size and(α=0.050) alpha level and95%confidence level(1-β) according to the power analysis. Each group consisted of 48 patients.

Randomizasyon Newborns meeting the inclusion criteria were randomly allocated to one of the 4 groups. Numbers were given to newborns sequentially on entry into the study and the random number stable used to allocate to one of 4 groups.

Physiological measurements Oxygen saturation Heart rate and oxygen saturations of newborns were examined using a pulse oximeter. A separate pulse oximetry probe was used for each baby.

Body temperature Newborns' body temperatures were measured using a non-contact thermometer. Bath water temperature The temperature of the water used for bathing was controlled using a bath thermometer.

Data Collection Tools The data were collected using the "Newborn Follow-up Form."

Newborn Follow-up Form:

This form was prepared by the researcher upon a literature review and included questions on the newborns' height, weight, diagnosis, gender, gestational age, physiological measurements (pulse, respiration, oxygen saturation, blood pressure, body temperature), and the delivery method.

PROCEDURE Preparation for applications The newborns' mothers were allowed to observe during the applications (massage, wipe bath and tub bath use). Suitable environmental conditions were provided for all newborns. The massages and wipe bathing were performed first by setting an appropriate temperature and humidity in the tub bathing . The door of the room used for bathing was kept closed, preventing heat loss and convection caused by air circulation. The room temperature and humidity were set to 26-28 °C and 40-60%, respectively. The duration of the applications was a maximum of 5 minutes. Clinical care of newborns (at least half an hour after feeding) and treatment processes were taken into consideration. In addition, the newborns were not touched until the evaluation was completed after the massage and bath.

For the massage application, alcohol-free and paraben-free baby oil with moisturising properties, suitable for newborns' skin type, was used. The temperature of the water used for the sponge bath was set at 37-38 °C, and separate cotton wipes were used for each body region. A folded cloth towel was placed in the tub bath before the bathing began. The water level inside the tub was set to 9-12 cm, deep enough to cover the newborn's shoulders. The temperature of the bath water was controlled using a special water thermometer.

The materials used during the applications were placed in easily accessible places, and nurses wore gloves after washing their hands prior to beginning the activities. All materials were disinfected after each application. The researchers were not involved in clinical follow-up of the infants, and nurses took all physiological measurements, recording them on the Newborn Follow-up Form.

Interventions Control Group The newborns in the control group did not undergo any intervention other than standard clinical practices. All physiological measurements (pulse, respiration, oxygen saturation and body temperature) were performed by nurses and recorded on the Newborn Follow-up Form.

Massage Group Massages were performed starting from the face, focused on the newborns forehead, and then around the eyes and cheeks with gentle touches. Then, newborns' chest area and the upper and lower extremities were massaged. Finally, newborns'were placed prone position and the back was massaged. Nurses recorded newborns' physiological measurements (pulse, respiration, oxygen saturation and body temperature) on the Newborn Follow-up Form.

Wipe Bathing Group In the sponge bathing group, the newborns' eyes, faces (outward from the midline), around the ear and the back of the ear were wiped from the inside out with cotton wipes and dried. Then, the chest area and arms, abdomen and back, legs and feet, respectively, were wiped and dried. Finally, the genital area was cleaned, before diapering the newborn. Nurses recorded newborns' physiological measurements (pulse, respiration, oxygen saturation and body temperature) on the Newborn Follow-up Form.

Tub Bathing Group In the tub bathing group, before being immersed in the tub, the newborns' faces and heads were cleaned outwards from the midline and dried. Then, the neck, chest, arms, back, legs and genital area were soaped, before the full body was rinsed and dried. Finally, umbilical cord care was performed, and the baby was diapered. Nurses recorded the newborns' physiological measurements (pulse, respiration, oxygen saturation and body temperature) on the Newborn Follow-up Form.

ELIGIBILITY:
Inclusion Criteria:

* newborns who born at 34 weeks' gestation and over
* newborns who receiving routine care and who were stable (temperature >36.5 °C, SpO2> 95%, HR = 120-160 / min)
* newborns who had an apgar score of 7 or higher at the first minute after birth;
* newborns who at least 24 hours old

Exclusion Criteria:

* newborns with any health problems that prevent bathing (eg congenital anomaly, surgical intervention, etc.)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-11-18 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in pulse | 30 minutes
  Nurses recorded the changes in pulse(HR) of newborns before, immediately after and 30 minutes after the intervention on the Newborn Follow up Survey.

SECONDARY OUTCOMES:
Changes in respiration | 30 minutes
  Nurses recorded the changes in respiration (O2) of newborns before, immediately after and 30 minutes after the intervention on the Newborn Follow up Survey.
:Changes in oxygen saturation | 30 minutes
  Nurses recorded the changes in oxygen saturation (SpO2) of newborns before, immediately after and 30 minutes after the intervention on the Newborn Follow up Survey.
Changes in body temperature | 30 minutes
  Nurses recorded the changes in body temperature (°C) of newborns before, immediately after and 30 minutes after the intervention on the Newborn Follow up Survey.

CONTACTS AND LOCATIONS:
Locations (1):
- Yeliz SUNA DAĞ, Malatya, Turkey (Türkiye)

REFERENCES:
- [Background] Loring C, Gregory K, Gargan B, LeBlanc V, Lundgren D, Reilly J, Stobo K, Walker C, Zaya C. Tub bathing improves thermoregulation of the late preterm infant. J Obstet Gynecol Neonatal Nurs. 2012 Mar;41(2):171-179. doi: 10.1111/j.1552-6909.2011.01332.x. Epub 2012 Feb 29. PMID 22375955
- [Result] Ala, H., Thaer, M., & Dina, S. (2010). The Effect of Timing of Initial Bath on Newborn's Temperature. Middle East Journal of Nursing, 4(3), 16-19.
- [Result] Ar I, Gozen D. Effects of Underrunning Water Bathing and Immersion Tub Bathing on Vital Signs of Newborn Infants: A Comparative Analysis. Adv Neonatal Care. 2018 Dec;18(6):E3-E12. doi: 10.1097/ANC.0000000000000484. PMID 30507829
- [Result] Association of Women's Health Obstetric and Neonatal Nurses, & (AWHONN). (2013). Neonatal skin care: Evidence-based clinical practice guideline. Washington: AWHONN
- [Result] Blume-Peytavi U, Lavender T, Jenerowicz D, Ryumina I, Stalder JF, Torrelo A, Cork MJ. Recommendations from a European Roundtable Meeting on Best Practice Healthy Infant Skin Care. Pediatr Dermatol. 2016 May;33(3):311-21. doi: 10.1111/pde.12819. Epub 2016 Feb 26. PMID 26919683
- [Result] Bryanton J, Walsh D, Barrett M, Gaudet D. Tub bathing versus traditional sponge bathing for the newborn. J Obstet Gynecol Neonatal Nurs. 2004 Nov-Dec;33(6):704-12. doi: 10.1177/0884217504270651. PMID 15561658
- [Result] Conk, Z., Başbakkal, Z., Bal Yılmaz, H., & Bolışık, B. (Eds.). (2013). Çocuk Sağlığı ve Hastalıkları Hemşireliği (Akademisye). Ankara.
- [Result] Caka SY, Gozen D. Effects of swaddled and traditional tub bathing methods on crying and physiological responses of newborns. J Spec Pediatr Nurs. 2018 Jan;23(1). doi: 10.1111/jspn.12202. Epub 2017 Nov 21. PMID 29160925
- [Result] Çavuşoğlu, H. (2013). Çocuk Sağlığı ve Hastalıkları Hemşireliği (Sistem Ofs). Ankara.
- [Result] Darmstadt GL, Dinulos JG. Neonatal skin care. Pediatr Clin North Am. 2000 Aug;47(4):757-82. doi: 10.1016/s0031-3955(05)70239-x. PMID 10943256
- [Result] Diego MA, Field T, Hernandez-Reif M. Vagal activity, gastric motility, and weight gain in massaged preterm neonates. J Pediatr. 2005 Jul;147(1):50-5. doi: 10.1016/j.jpeds.2005.02.023. PMID 16027695
- [Result] Diego MA, Field T, Hernandez-Reif M. Temperature increases in preterm infants during massage therapy. Infant Behav Dev. 2008 Jan;31(1):149-52. doi: 10.1016/j.infbeh.2007.07.002. Epub 2007 Aug 9. PMID 17692385
- [Result] Jain S, Kumar P, McMillan DD. Prior leg massage decreases pain responses to heel stick in preterm babies. J Paediatr Child Health. 2006 Sep;42(9):505-8. doi: 10.1111/j.1440-1754.2006.00912.x. PMID 16925535
- [Result] Kurtulan Bulut, H. (2009). Prematüre Bebeklerde İki Banyo Yönteminin Fizyolojik Ölçüm Sonuçlarına Etkisi. Dokuz Eylül Üniversitesi.
- [Result] Lee HK. Effects of sponge bathing on vagal tone and behavioural responses in premature infants. J Clin Nurs. 2002 Jul;11(4):510-9. doi: 10.1046/j.1365-2702.2002.00594.x. PMID 12100647
- [Result] Lin CH, Yang HC, Cheng CS, Yen CE. Effects of infant massage on jaundiced neonates undergoing phototherapy. Ital J Pediatr. 2015 Nov 25;41:94. doi: 10.1186/s13052-015-0202-y. PMID 26607061
- [Result] Mangalgi, S., & Upadhya, N. (2014). Variation of Body Temperature After Sponge Bath in Stable Very Low Birth Weight Preterm Neonates. Indian J Child Health, 4(2), 221-224. https://doi.org/10.4158/EP13328.OR
- [Result] Medves JM, O'Brien B. The effect of bather and location of first bath on maintaining thermal stability in newborns. J Obstet Gynecol Neonatal Nurs. 2004 Mar-Apr;33(2):175-82. doi: 10.1177/0884217504263081. PMID 15095796
- [Result] Morelius E, Hellstrom-Westas L, Carlen C, Norman E, Nelson N. Is a nappy change stressful to neonates? Early Hum Dev. 2006 Oct;82(10):669-76. doi: 10.1016/j.earlhumdev.2005.12.013. Epub 2006 Feb 28. PMID 16507341
- [Result] Smith SL, Haley S, Slater H, Moyer-Mileur LJ. Heart rate variability during caregiving and sleep after massage therapy in preterm infants. Early Hum Dev. 2013 Aug;89(8):525-9. doi: 10.1016/j.earlhumdev.2013.01.004. Epub 2013 Jan 27. PMID 23361061
- [Result] Sülü Uğurlu, E. (2011). Aşı Uygulanan Bebeklerde Ağrının Giderilmesinde Bacak Masajının Etkisinin İncelenmesi. Dokuz Eylül Üniversitesi.
- [Result] Tasdemir HI, Efe E. The effect of tub bathing and sponge bathing on neonatal comfort and physiological parameters in late preterm infants: A randomized controlled trial. Int J Nurs Stud. 2019 Nov;99:103377. doi: 10.1016/j.ijnurstu.2019.06.008. Epub 2019 Jun 21. PMID 31442786
- [Result] Törüner, E. ., & Lale, B. (2011). Çocuk sağlığı: temel hemşirelik yaklaşımları (Göktuğ yay). Ankara.
- [Result] Varda KE, Behnke RS. The effect of timing of initial bath on newborn's temperature. J Obstet Gynecol Neonatal Nurs. 2000 Jan-Feb;29(1):27-32. doi: 10.1111/j.1552-6909.2000.tb02753.x. PMID 10660274
- [Result] Yıldız, S. (2008). İlk günden sonraki bakım. İçinde: Temel neonatoloji ve hemşirelik ilkeleri. (T. Dağoğlu & G. Görak, Eds.) (Nobel Tıp). İstanbul.